CLINICAL TRIAL: NCT03539848
Title: The Use of a Portable 3D Head Mounted Display (HMD) With Integrated Eye Capture Technology (IPAS Goggles) for the Diagnosis of Mild Traumatic Brain Injury (mTBI) in a Community Setting
Brief Title: Diagnosis of mTBI in a Community Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Neurolign (Industry)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20180012
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury; Brain Injuries; Brain Injuries, Traumatic; Head Injury
Keywords: TBI; Community Setting; Mild TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Brain Injuries; Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subjects with mTBI (Experimental): Individuals who come to the emergency department or urgent/acute care facility with an mTBI will undergo testing with the I-PAS Goggles.
  Interventions: Device: I-PAS Goggles
- Subjects with minor injuries (Active Comparator): Individuals who come to the emergency department or urgent/acute care facility with minor injuries (such as ankle sprains or knee sprains) will undergo testing with the I-PAS Goggles.
  Interventions: Device: I-PAS Goggles

INTERVENTIONS:
Device: I-PAS Goggles — Portable, head-mounted display goggle system with integrated eye capture technology

SUMMARY:
The purpose of this research study is to test whether a portable goggle system (I-PAS) is good at diagnosing mild traumatic brain injury (mTBI) in a community setting. The goal is to determine whether the IPAS goggle system can be used reliably in an urgent care or emergency department setting.

DETAILED DESCRIPTION:
The purpose of this research study is to test whether a portable goggle system (I-PAS) is good at diagnosing mild traumatic brain injury (mTBI) in a community setting. The goal is to determine whether the IPAS goggle system can be used reliably in an urgent care or emergency department setting. The study further looks at current metrics and compares their efficacy in both the diagnosis and prognostic value of individuals with mTBI.

ELIGIBILITY:
Participants must meet one of the following inclusion criteria:

1. Males and females from 18-50 years of age who present to the emergency department or urgent/acute care facility at the University of Miami Hospital, Jackson Memorial Hospital, or by direct referral to the clinic with a history of all of the following: 1) Blow or impact to head, 2) Period of loss or alteration of consciousness, 3) Neurosensory symptoms, and 4) Diagnosis by Emergency Room Staff or Medical Staff of having suffered an mTBI/Concussion.
2. An age- and sex- matched control group also recruited from emergency department or urgent/acute care facility at the University of Miami Hospital, Jackson Memorial Hospital, or by direct referral to the clinic. These will include individuals with minor injuries (e.g ankle sprains, minor knee injuries, etc.) not involving the head and not requiring admission to the hospital.

Exclusion Criteria:

1. History of head injury characterized by any of the following:

   1. Resulting from penetrating trauma
   2. Resulting from an automobile accident with significant associated injuries
   3. Associated with a Glasgow Comma Scale Score of less than 13 at the time of injury
   4. Associated with a loss of consciousness period greater than 59 minutes
   5. Judged to be more than mild by Medical Staff
   6. Requiring admission to the hospital for any reason
   7. Associated with subdural or epidural hemorrhage
2. Head injury history

   1. For control group - history of head injury within the last six months or currently experience any head injury symptoms at time of enrollment
   2. For head injured group - history of head injury within the last three months or experiencing head injury symptoms immediately prior to the current head injury
3. Presence of severe aphasia
4. History of diagnosed neuropsychiatric disorders (e.g. hypochondriasis, major depression, schizophrenia)
5. Documented neurodegenerative disorders
6. Pregnancy [Female candidates will be asked if they are pregnant]
7. Prior disorders of hearing and balance including:

   1. Meniere's disease
   2. Multiple sclerosis
   3. Vestibular neuritis
   4. Vestibular schwannoma
   5. Sudden sensorineural hearing loss
8. History of Cerebrovascular disorders
9. History of ear operation other than myringotomy and tube placement in the past
10. Systemic disorders to include chronic renal failure, cirrhosis of the liver, autoimmune disease, heart disease, lung disease, or severe arthritis
11. Children
12. Individuals who cannot provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with mTBI | 33 months
  How many participants were detected to have mTBI following an injury.

SECONDARY OUTCOMES:
Time to recover | 33 months
  Measuring the time (days) it takes for readiness to return to normal activity after a head injury for participants with a detected mTBI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoffer, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No